CLINICAL TRIAL: NCT02341105
Title: AMIOCAAF (AMIOdarone vs. Catheter Ablation for Prevention of Recurrent Symptomatic Atrial Fibrillation): a Randomized Controlled Trial - Vanguard Phase
Brief Title: AMIOdarone vs. Catheter Ablation for Prevention of Recurrent Symptomatic Atrial Fibrillation
Acronym: AmioCAAF
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: low recruitment rate
Sponsor: Population Health Research Institute (Other)
Collaborators: Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AmioCaAF1
Record Dates: First submitted 2015-01-11; First posted 2015-01-19 (Estimated); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation; Amiodarone; Anti-Arrhythmia Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Medical therapy (Active Comparator): Amiodarone treatment. Amiodarone will be given at a loading dose of 400 mg per day for two week and then lowered to 200 mg daily for 6 months at which point the dose will be lowered to 1000 mg per week. The dose of amiodarone will then be lowered every six, as long as the patient has a satisfactory response. The minimum dose will be 700 mg per week.
  Interventions: Drug: Amiodarone
- Catheter ablation (Active Comparator): A standard pulmonary vein isolation procedure will be done. Additional ablation will be permitted (roof and mitral lines/ CFAE )
  Interventions: Procedure: Catheter ablation

INTERVENTIONS:
Procedure: Catheter ablation — Pulmonary vein isolation by catheter ablation
  Other Names: Pulmonary Vein Isolation (PVI)
  Arms: Catheter ablation
Drug: Amiodarone — antiarrhythmic therapy using Amiodarone
  Other Names: Antiarrhythmic
  Arms: Medical therapy

SUMMARY:
Randomized trial of low-dose amiodarone therapy versus catheter ablation (CA) in older patients with persistent atrial fibrillation (AF).

Primary Objective: To compare amiodarone to catheter ablation in patients aged 50 to 80 years with symptomatic AF for the composite outcome of hospitalization for cardiovascular cause or emergency department visit for atrial arrhythmia

DETAILED DESCRIPTION:
This is a single centre vanguard phase prospective randomized open label study with blinded outcome adjudication.

Patients will be randomized by a central randomization system (1:1) to amiodarone or catheter ablation.

1. Amiodarone will be started at a dose of 400 mg/day. After one month the dose will be lowered to 200 mg per day. Patients will be seen every six months. At each visit the dose of amiodarone will be lowered by 100 mg per week if the patient is having a good clinical response to treatment. Good clinical response will be a a clinical assessment that takes into account not only actual or possible arrhythmia recurrence but also side-effects and patient acceptability of treatment. A minimum dose of 700 mg/week will be allowed. If patient symptoms recur, the amiodarone dose may be increased but not above a dose of 200 mg/day .
2. Catheter ablation of persistent AF will be done within two months using pulmonary vein isolation in all subjects
3. Patient not in sinus rhythm at time randomization will undergo DC cardioversion after at least 1 month of amiodarone Rx or during CA.

Follow up: Clinical assessment will include a medical history and physical examination to be performed at baseline, and every 3 months. This will also include 12-lead ECG.

b. At 3, 6, 12, 18, and 24 months: QOL questionnaire (AFEQT- Atrial Fibrillation Effect on QualiTy of life) c. Thyroid and liver function tests, chest X-ray will be obtained at regular intervals.

d. Arrhythmia will be monitored using a 2-week event monitors at 6, 12, 18, 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Recurrent symptomatic Atrial Fibrillation (AF)
2. Age 50-80 years with persistent AF (≥1 of AF episode lasting more than a week or requiring cardioversion)

Exclusion Criteria:

1. Permanent atrial fibrillation
2. Prior continuous use of amiodarone of more than 2 weeks.
3. Prior catheter ablation for AF.
4. Have a documented resting heart (while awake) of < 50 beats per minute.
5. Have a known severe liver disease.
6. Are deemed not suitable for CA (LA size, comorbidities…).
7. Have a severe valvular disease or have a mechanical mitral prosthesis.
8. Have a life-expectancy of less than 2 years.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-01; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
The composite outcome of hospitalization for cardiovascular cause or emergency department visit for atrial arrhythmia. | 2 years

SECONDARY OUTCOMES:
First recurrence of an atrial tachyarrhythmia documented on 12 lead ECG or a 14-day event monitor | 2 years
First recurrence of a symptomatic atrial tachyarrhythmia documented on 12 lead ECG or a 14-day event monitor | 2 years
Quality of life measured at 3, 6 and 12 months using the Atrial Fibrillation Effect on QualiTy of Life Survey (AFEQT) | 2 years

OTHER OUTCOMES:
Potential Side Effects Related to amiodarone or ablation procedure | 2 years
  Known potential side effects of catheter ablation include vascular access complications such as hematoma, pseudoaneurysm, or AV fistula. Less common but more serious include cardiac perforation (0.5%-1%) and thromboembolism (0.5%-1%), and fatal complications occur in approximately 1:1000 cases.
  Known potential side effects of amiodarone include amiodarone toxicity, corneal micro-deposits, photosensitivity, thyroid abnormalities. pulmonary toxicity, abnormal liver function, and skin discolouration.

CONTACTS AND LOCATIONS:
Overall Officials: Guy Amit, MD, Principal Investigator — Hamilton Heath Sciences
Locations (1):
- Hamilton Health Sciences, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No